CLINICAL TRIAL: NCT07354724
Title: A Phase 1, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL952 in Adult Participants With Late-Onset Pompe Disease
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of DNL952 in Adult Participants With Late-Onset Pompe Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DNLI-J-0001; 2025-524082-25-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Late-onset Pompe Disease
Keywords: LOPD; Pompe; acid maltase deficiency; glycogen storage disease type II; ERT; enzyme replacement therapy
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A1 (Experimental): Participants with LOPD
  Interventions: Drug: DNL952
- Cohort A2 (Experimental): Participants with LOPD
  Interventions: Drug: DNL952
- Cohort A3 (Optional) (Experimental): Participants with LOPD
  Interventions: Drug: DNL952
- Cohort A4 (Optional) (Experimental): Participants with LOPD
  Interventions: Drug: DNL952
- Cohort B1 (Optional) (Experimental): Participants with LOPD
  Interventions: Drug: DNL952
- Cohort B2 (Optional) (Experimental): Participants with LOPD
  Interventions: Drug: DNL952

INTERVENTIONS:
Drug: DNL952 — Intravenous repeating dose

SUMMARY:
This is a Phase 1, multicenter, open-label study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of DNL952 in adult participants with late-onset Pompe disease. The principal aim of this study is to obtain safety and tolerability data across varous dose levels of DNL952 in participants with late-onset Pompe disease (LOPD).

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight ≥40 kg
* Diagnosis of LOPD
* Upright FVC ≥ 30% of predicted normal value
* Able to ambulate ≥ 40 meters (use of assistive devices is acceptable)
* [Cohorts A1-A4 only] Have received avalglucosidase alfa or cipaglucosidase alfa at a dose of 20 mg/kg every 2 weeks for at least 12 months prior to screening
* [Cohorts B1-B2 only] Must not have received any enzyme-replacement therapy for Pompe disease in the 12 months prior to screening

Key Exclusion Criteria:

* Any ongoing, clinically significant, unstable, or poorly controlled neurological, psychiatric, endocrine, pulmonary, cardiovascular, gastrointestinal, hepatic, pancreatic, renal, metabolic, hematological, immunological, allergic, or ophthalmic disease not related to Pompe disease, or other major disorders. Well-controlled conditions are permitted if investigator and Sponsor agree.
* Wheelchair-dependent
* Require noninvasive ventilation for an average of more than 6 hours per day while awake or any invasive ventilation. Use of noninvasive ventilation during sleep is acceptable.
* Received an experimental gene therapy at any time or participation in any other investigational drug trial or use of investigational drug within 60 days or 5 half-lives, whichever is longer, before screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and seriousness of treatment-emergent adverse events (TEAEs) | 48 weeks
Incidence and severity of infusion-related reacations (IRRs) | 48 weeks

SECONDARY OUTCOMES:
PK parameter: Maximum concentration (Cmax) of DNL952 in serum | 48 weeks
PK Parameter: Time to reach maximum concentration (tmax) of DNL952 in serum | 48 weeks
PK Parameter: Area under the concentration-time curve (AUC) from time zero to time of last measurable concentration (AUClast) of DNL952 in serum | 48 weeks
PK Parameter: AUC from time 0 to infinity (AUC∞) of DNL952 in serum | 48 weeks
  single dose only
PK parameter: AUC from time zero to time t (AUCt) of DNL952 in serum | 48 weeks
  multiple doses only
PK Parameter: terminal elimination half-life (t1/2) of DNL952 in serum | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Denali Therapeutics Inc.

IPD SHARING:
Plan to Share IPD: No